CLINICAL TRIAL: NCT01236534
Title: Single-center, Randomized, Double-blind, Placebo-controlled, Parallel-groups Study of Lubiprostone in Patients With Multiple Sclerosis-Associated Constipation
Brief Title: Lubiprostone in Patients With Multiple Sclerosis Associated Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Andrew Goodman, MD, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URMC08-022LUB
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Sclerosis; Constipation
Keywords: Multiple Sclerosis; Constipation; Multiple Sclerosis Associated Constipation
MeSH Terms: conditions — Multiple Sclerosis; Constipation | interventions — Lubiprostone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone (Active Comparator)
  Interventions: Drug: Lubiprostone
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — 24 mcg twice daily for 21 days.
  Other Names: Amitiza
  Arms: Lubiprostone
Drug: Placebo — matching placebo twice daily for 21 days.
  Other Names: Sugar pill
  Arms: Sugar pill

SUMMARY:
The purpose of the study is to assess how safe and effective the drug Lubiprostone is in people with Multiple Sclerosis (MS)and moderate to severe MS-associated constipation. Lubiprostone is approved by the FDA for the treatment of two common types of constipation in adults, chronic idiopathic constipation and irritable bowel syndrome.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a disorder of the body's immune system that affects the central nervous system. Normally, nerve fibers carry electrical impulses through the spinal cord, providing communication between the brain and the bowel. In people with MS, the covering around the nerve fibers deteriorates, causing nerve impulses to be slowed or stopped. as a result, patients with MS may experiences constipation.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis
* Chronic Constipation defined as < 3 spontaneous bowel movements per week by history and confirmed by diary during the 14 day washout period.
* Women of child-bearing potential must agree to use adequate birth control.

Exclusion Criteria:

* history of other clinically significant medical or psychiatric disorders or suicidal ideation.
* Subjects who have a suspicion of a mechanical bowel obstruction by clinical evaluation prior to dosing that include nausea, vomiting, abdominal pain or distention.
* Subjects with a positive urine pregnancy test prior to dosing.
* Medication changes within one month prior to visit one.
* Corticosteroid use within 2 months prior to visit one.
* Age<18.
* Known intolerance to lubiprostone.
* Inability to perform any required study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Goodman, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured in the Multiple Sclerosis Clinic at the University of Rochester, which began on 08/30/2010 until the last subject was enrolled on 12/27/2011.
Pre-assignment Details: After inclusion criteria and screening, subjects were instructed to D/C all over the counter and Rx bowel medications except for fiber supplements for 14 days. Any subject with >2 BM/Week were excluded. 40 patients screened and 21 randomization, 18 were ineligible D/T a high baseline SBM count, and 1 was unable to reschedule.
Groups:
- Lubiprostone: Lubiprostone : 24 mcg twice daily for 21 days.
- Sugar Pill: Placebo : matching placebo twice daily for 21 days.
Period: Overall Study
Arm/Group | Lubiprostone | Sugar Pill
Started | 11 | 10
Completed | 8 (2 subjects stopped treatment due to diarrhea, and 1 stopped treatment due to constipation.) | 10
Not Completed | 3 | 0
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubiprostone | Sugar Pill | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (14.8) | 41.6 (8.8) | 44.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Spontaneous Bowel Movements in Patients With Multiple Sclerosis (MS)-Associated Constipation Per Day.
Description: Number of of lubiprostone 24 mcg twice daily on spontaneous bowel movements (SBM) in patients with multiple sclerosis (MS)-associated constipation per day. Hypothesis: Lubiprostone-treated patients will have more SBM's than placebo-treated patients.
Time Frame: 21 days
Population: per protocol
Measure: Mean (Standard Deviation); unit: spontaneous bowel movements
Arm/Group | Lubiprostone | Sugar Pill
Number analyzed (Participants) | 11 | 10
spontaneous bowel movements | 3.4 (0.7) | 3.2 (0.6)

2. Secondary Outcome: Number of Participants With Diarrheic Events.
Description: To determine the safety of lubiprostone based on adverse event (AE) type, frequency, and severity. Hypothesis: AE type, frequency, and severity will be comparable in lubiprostone and placebo treated patients.
Time Frame: 21 days
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Lubiprostone | Sugar Pill
Number analyzed (Participants) | 11 | 10
participants | 8 | 2

ADVERSE EVENTS:
Arm/Group | Lubiprostone | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 8/11 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubiprostone (N=11) | Sugar Pill (N=10)
diarrhea (Gastrointestinal disorders) | 8 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less